CLINICAL TRIAL: NCT01627912
Title: Acute Effects of Wine Consumption on Platelet Aggregation, and on Inflammatory / Oxidative Stress Markers
Brief Title: Acute Effects of Wine Consumption on Healthy Volunteers
Acronym: winepost
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Harokopio University (Other)
Collaborators: Graduate Program of the Department of Nutrition and Dietetics (Unknown)
Responsible Party: Principal Investigator, Elizabeth Fragopoulou, PhD, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HUABIO01
Record Dates: First submitted 2012-06-14; First posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Healthy, Postprandial
Keywords: wine; inflammation; oxidative stress; randomized control trial; postprandial intervention; platelet aggregation; haemostasis; robola; cabernet sauvignon; alcohol; PAF metabolism
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Robola, Cabernet Sauvignon wines — 4 treatments on separate days: the subjects randomly consumed 4ml of drink [white wine or red wine or 12.5% ethanol or water]/kg of individual, parallel with a standardized meal.

SUMMARY:
The purpose of this study is to investigate whether red and white wine consumption has acute effects on postprandial biochemical markers related to platelet aggregation, inflammation and oxidative stress compared to water or 12.5% ethanol aqueous solution consumption.

DETAILED DESCRIPTION:
The last few years, epidemiologic studies indicate that regular moderate consumption of alcohol is associated with lower risk of coronary heart disease and heart attack, as well as with lower mortality. More specific, a J or U-shaped association between alcohol consumption and the incidence of coronary heart disease have been suggested, which means that there was lower disease risk in moderate alcohol consumers than in abstainers or heavy drinkers.

The scientific interest was focused on wine after the term "French paradox" was introduced, in order to describe the epidemiological observation that the French suffer a relatively low incidence of coronary heart disease, despite having a diet relatively rich in saturated fats. The paradox was attributed to the moderate consumption of red wine by French. Even though many clinical studies have occurred since then, only few of them report the postprandial effect of wine, mainly focusing on the study of oxidative stress markers and endothelium dysfunction. Also, a limited number of publications refer to the postprandial wine effect upon platelet aggregation, which is an indicative marker for inflammation / thrombosis and atherosclerosis.

The limited clinical evidence prompted us to investigate the postprandial effect of wine consumption upon platelet aggregation, inflammation and oxidation markers, by undertaking a clinical study of crossover design. The subjects randomly consumed 4ml of drink [Robola or Cabernet Sauvignon or 12.5% ethanol or water]/kg of individual, parallel with a standardized meal, which consisted of 30.8% carbohydrates, 12.0% proteins and 53.1% fat. The meal total energy was 787.2 kcal.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-obese

Exclusion Criteria:

* smokers
* those who reported slimming or any other dietary regime
* abstainers from alcohol consumption
* heavy drinkers
* athletes
* subjects who were on medication, such as aspirin, that may have an impact on platelet aggregation or surgical events that may have affected the study outcomes
* participants with a known diagnosis of either hypertension or diabetes
* subjects on medication

Ages: 26 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
platelet aggregation | baseline
  In each time point platelet rich plasma (PRP) was isolated from the blood of volunteers and platelet aggregation upon Platelet activating factor (PAF) was measured in CHRONO-LOG aggregometer.
platelet aggregation | 30 min after standardized meal plus tested drink consumption.
  In each time point platelet rich plasma (PRP) was isolated from the blood of volunteers and platelet aggregation upon Platelet activating factor (PAF) was measured in CHRONO-LOG aggregometer.
platelet aggregation | 90 min after standardized meal plus tested drink consumption.
  In each time point platelet rich plasma (PRP) was isolated from the blood of volunteers and platelet aggregation upon Platelet activating factor (PAF) was measured in CHRONO-LOG aggregometer.
platelet aggregation | 150 min after standardized meal plus tested drink consumption
  In each time point platelet rich plasma (PRP) was isolated from the blood of volunteers and platelet aggregation upon Platelet activating factor (PAF) was measured in CHRONO-LOG aggregometer.
platelet aggregation | 210 min after standardized meal plus tested drink consumption.
  In each time point platelet rich plasma (PRP) was isolated from the blood of volunteers and platelet aggregation upon Platelet activating factor (PAF) was measured in CHRONO-LOG aggregometer.
platelet aggregation | 300 min after standardized meal plus tested drink consumption.
  In each time point platelet rich plasma (PRP) was isolated from the blood of volunteers and platelet aggregation upon Platelet activating factor (PAF) was measured in CHRONO-LOG aggregometer.
markers of inflammation | baseline
markers of inflammation | 0 min after standardized meal plus tested drink consumption
markers of inflammation | 30 min after standardized meal plus tested drink consumption
markers of inflammation | 60 min after standardized meal plus tested drink consumption
markers of inflammation | 90 min after standardized meal plus tested drink consumption
markers of inflammation | 120 min after standardized meal plus tested drink consumption
markers of inflammation | 150 min after standardized meal plus tested drink consumption
markers of inflammation | 180 min after standardized meal plus tested drink consumption
markers of inflammation | 210 min after standardized meal plus tested drink consumption
markers of inflammation | 240 min after standardized meal plus tested drink consumption
markers of inflammation | 300 min after standardized meal plus tested drink consumption
markers of inflammation | 360 min after standardized meal plus tested drink consumption
markers of oxidative stress | baseline
  TBARS, ex vivo serum oxidation etc
markers of oxidative stress | 0 min after standardized meal plus tested drink consumption
  TBARS, ex vivo serum oxidation etc
markers of oxidative stress | 30 min after standardized meal plus tested drink consumption
  TBARS, ex vivo serum oxidation etc
markers of oxidative stress | 60 min after standardized meal plus tested drink consumption
  TBARS, ex vivo serum oxidation etc
markers of oxidative stress | 90 min after standardized meal plus tested drink consumption
  TBARS, ex vivo serum oxidation etc
markers of oxidative stress | 120 min after standardized meal plus tested drink consumption
  TBARS, ex vivo serum oxidation etc
markers of oxidative stress | 150 min after standardized meal plus tested drink consumption
  TBARS, ex vivo serum oxidation etc
markers of oxidative stress | 180 min after standardized meal plus tested drink consumption
  TBARS, ex vivo serum oxidation etc
markers of oxidative stress | 210 min after standardized meal plus tested drink consumption
  TBARS, ex vivo serum oxidation etc
markers of oxidative stress | 240 min after standardized meal plus tested drink consumption
  TBARS, ex vivo serum oxidation etc
markers of oxidative stress | 300 min after standardized meal plus tested drink consumption
  TBARS, ex vivo serum oxidation etc
markers of oxidative stress | 360 min after standardized meal plus tested drink consumption
  TBARS, ex vivo serum oxidation etc
PAF metabolism | 0 min after standardized meal plus tested drink consumption
  Measurement of PAF biosynthetic / catabolic enzymes in leucocytes and LpPLA2 in serum
PAF metabolism | 60 min after standardized meal plus tested drink consumption
  Measurement of PAF biosynthetic / catabolic enzymes in leucocytes and LpPLA2 in serum
PAF metabolism | 90 min after standardized meal plus tested drink consumption
  Measurement of PAF biosynthetic / catabolic enzymes in leucocytes and LpPLA2 in serum
PAF metabolism | 120 min after standardized meal plus tested drink consumption
  Measurement of PAF biosynthetic / catabolic enzymes in leucocytes and LpPLA2 in serum
PAF metabolism | 180 min after standardized meal plus tested drink consumption
  Measurement of PAF biosynthetic / catabolic enzymes in leucocytes and LpPLA2 in serum
PAF metabolism | 210 min after standardized meal plus tested drink consumption
  Measurement of PAF biosynthetic / catabolic enzymes in leucocytes and LpPLA2 in serum
PAF metabolism | 240 min after standardized meal plus tested drink consumption
  Measurement of PAF biosynthetic / catabolic enzymes in leucocytes and LpPLA2 in serum
PAF metabolism | 300 min after standardized meal plus tested drink consumption
  Measurement of PAF biosynthetic / catabolic enzymes in leucocytes and LpPLA2 in serum
PAF metabolism | 360 min after standardized meal plus tested drink consumption
  Measurement of PAF biosynthetic / catabolic enzymes in leucocytes and LpPLA2 in serum

SECONDARY OUTCOMES:
Glucose levels | baseline
Glucose levels | 0 min after standardized meal plus tested drink consumption
Glucose levels | 30 min after standardized meal plus tested drink consumption
Glucose levels | 60 min after standardized meal plus tested drink consumption
Glucose levels | 90 min after standardized meal plus tested drink consumption
Glucose levels | 120 min after standardized meal plus tested drink consumption
Glucose levels | 150 min after standardized meal plus tested drink consumption
Glucose levels | 180 min after standardized meal plus tested drink consumption
Glucose levels | 210 min after standardized meal plus tested drink consumption
Glucose levels | 240 min after standardized meal plus tested drink consumption
Glucose levels | 300 min after standardized meal plus tested drink consumption
Glucose levels | 360 min after standardized meal plus tested drink consumption
Insulin levels | 0 min after standardized meal plus tested drink consumption
Insulin levels | 30 min after standardized meal plus tested drink consumption
Insulin levels | 60 min after standardized meal plus tested drink consumption
Insulin levels | 90 min after standardized meal plus tested drink consumption
Insulin levels | 120 min after standardized meal plus tested drink consumption
lipids | baseline
  HDL-cholesterol, LDL-cholesterol, total chlesterol, triglycerides
lipids | 0 min after standardized meal plus tested drink consumption
  HDL-cholesterol, LDL-cholesterol, total chlesterol, triglycerides
lipids | 30 min after standardized meal plus tested drink consumption
  HDL-cholesterol, LDL-cholesterol, total chlesterol, triglycerides
lipids | 60 min after standardized meal plus tested drink consumption
  HDL-cholesterol, LDL-cholesterol, total chlesterol, triglycerides
lipids | 90 min after standardized meal plus tested drink consumption
  HDL-cholesterol, LDL-cholesterol, total chlesterol, triglycerides
lipids | 120 min after standardized meal plus tested drink consumption
  HDL-cholesterol, LDL-cholesterol, total chlesterol, triglycerides
lipids | 150 min after standardized meal plus tested drink consumption
  HDL-cholesterol, LDL-cholesterol, total chlesterol, triglycerides
lipids | 180 min after standardized meal plus tested drink consumption
  HDL-cholesterol, LDL-cholesterol, total chlesterol, triglycerides
lipids | 210 min after standardized meal plus tested drink consumption
  HDL-cholesterol, LDL-cholesterol, total chlesterol, triglycerides
lipids | 240 min after standardized meal plus tested drink consumption
  HDL-cholesterol, LDL-cholesterol, total chlesterol, triglycerides
lipids | 300 min after standardized meal plus tested drink consumption
  HDL-cholesterol, LDL-cholesterol, total chlesterol, triglycerides
lipids | 360 min after standardized meal plus tested drink consumption
  HDL-cholesterol, LDL-cholesterol, total chlesterol, triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Fragopoulou, Chemist PhD, Principal Investigator — Department of Nutrition-Dietetics, Harokopio University, Athens, Greece
Locations (1):
- Department of Nutrition-Dietetics, Harokopio University, Athens, Greece